CLINICAL TRIAL: NCT00915837
Title: Phase 1 Prospective, Randomized, Double-Masked, Multicenter Study to Evaluate the Safety and Tolerability of Two Dose Levels of the Helical Intravitreal Triamcinolone Implant in Diabetic Macular Edema
Brief Title: Safety and Tolerability Study of the Helical Intravitreal Triamcinolone Implant in Diabetic Macular Edema
Acronym: STRIDE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRDX- 001
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2009-06

CONDITIONS: Diabetic Macular Edema
Keywords: DME
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow release formulation (Experimental): Slow release formulation, helical intravitreal triamcinolone implant
  Interventions: Drug: triamcinolone acetonide
- fast release formulation (Experimental): fast release formulation, helical intravitreal triamcinolone implant
  Interventions: Drug: triamcinolone acetonide

INTERVENTIONS:
Drug: triamcinolone acetonide — Helical intravitreal triamcinolone implant- 925 mcg drug; slow release formulation approximately 1-3 mcg/day
  Arms: Slow release formulation
Drug: triamcinolone acetonide — Helical intravitreal triamcinolone implant- 925 mcg drug; fast release formulation approximately 3-5 mcg/day
  Arms: fast release formulation

SUMMARY:
This Phase 1 study will evaluate the safety, tolerability and duration of effect of a helical intravitreal triamcinolone implant for the treatment of diabetic macular edema over a three-year period.

DETAILED DESCRIPTION:
The Helical Intravitreal Triamcinolone Implant is intended to provide sustained release of triamcinolone acetonide into the vitreous chamber of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically observable macular edema associated with diabetic retinopathy in study eye
* Macular edema in study eye is associated with

  1. visual acuity of 20/40 or worse; and
  2. retinal thickening in the fovea as seen on biomicroscopic examination
  3. angiographic evidence of leakage involving the perifoveal capillary net
* Failure of macular edema to improve with prior macular photocoagulation, or the patient is unlikely to benefit from macular photocoagulation in the opinion of the investigator
* Patients must be 18 years of age and older
* Patients must be willing and able to return for scheduled follow up examinations for 3 years after initial surgery.
* Patients must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Monocular, or vision worse than 20/400 in the fellow eye
* Visual acuity worse than 20/200 20/200 and < 34 letters read in the study eye
* Use of depot periocular steroids in the study eye within the past 30 days
* Current use of >15 mg/day of oral steroids
* Known steroid responder
* Ocular hypertension > 22 mmHg in the study eye or need for more than one medication to maintain IOP < 22 mmHg.
* Cup to disc ratio of > 0.8 in the study eye
* Prior filtration surgery or glaucoma implant surgery in the study eye
* Any active ocular infection in either eye
* History of herpetic ocular infection in the study eye
* Macular ischemia, defined as angiographic evidence of enlargement of the foveal avascular zone to 1 disc area or larger, centered on the fovea
* Macular or panretinal photocoagulation treatment in the study eye within the past 90 days; laser capsulotomy within the past 90 days
* Planned or known need for ocular surgery in the study eye within 90 days after enrollment and treatment
* Any condition that precludes the subject's ability to comply with study requirements, including examinations or the completion of the study; or any condition that precludes the examiner's ability to obtain reliable fundus photography, angiography, or OCT images
* Females who are pregnant or lactating, and premenopausal females who are unwilling to use a medically accepted method of birth control for the duration of the study
* Participation in another investigational trial within 30 days prior to enrollment or during the study period
* Uncontrolled hypertension (systolic BP > 160 mm Hg and/or diastolic BP > 90 mmHg)
* Uncontrolled diabetes (HbA1c > 13)
* Chronic renal failure requiring dialysis or anticipated renal transplant
* Retinal or choroidal neovascularization in the study eye; anticipated need for panretinal photocoagulation within the next 30 days
* Macular edema in the study eye known to be due to a cause other than diabetic retinopathy
* Use of immunosuppressant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-06; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | every 3 months for 36 months

SECONDARY OUTCOMES:
OCT | every 3 months for 36 months
IOP | every 3 months for 36 months
Slit lamp exam/funduscopy | every 3 months for 36 months
Fluorescein angiography | every 3 months for 36 months
Adverse events | every 3 months for 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L Cantrill, MD, Principal Investigator — VitreoRetinal Surgery, PA; Pravin U Dugel, MD, Principal Investigator — Retinal Consultants of Arizona; Tamer H Mahmoud, MD, PhD, Principal Investigator — Kresege Eye Institute; Robert L Avery, MD, Principal Investigator — California Retinal Consultants
Locations (4):
- United States (4):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Santa Barbara, California
  - Kresege Eye Institute, Detroit, Michigan
  - VitreoRetinal Surgery, PA, Edina, Minnesota